CLINICAL TRIAL: NCT00794872
Title: Hyperoxic Chemoreflex Sensitivity in Chronic Kidney Disease
Brief Title: Chemoreflex Sensitivity in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other); SLK Kliniken Heilbronn GmbH (Other)
Responsible Party: Christian Meyer, MD, RWTH Aachen University
Other Study IDs: Chemoreflex-Sensitivity-Study
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Kidney Disease; Cardiovascular Morbidity
Keywords: Cardiovascular autonomic neuropathy; Chemoreflex sensitivity; Chronic kidney disease; Sudden cardiac arrest
MeSH Terms: conditions — Renal Insufficiency, Chronic; Death, Sudden, Cardiac | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Measurement of the venous partial pressure of oxygen in blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Patients with stage 3 CKD
  Interventions: Other: blood sampling
- 2: Patients with stage 4 CKD
  Interventions: Other: blood sampling
- 3: Patients without evidence for CDK
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling

SUMMARY:
Cardiovascular morbidity and mortality are markedly increased in chronic kidney disease (CKD) and may be explained in part by sympathetic hyperactivity. Impaired hyperoxic chemoreflex sensitivity (CHRS) has been attributed to an increased sympathetic activity. The aim of the present study is to examine whether chemosensor function is altered in patients with stage 3 and stage 4 CKD.

DETAILED DESCRIPTION:
Impaired hyperoxic chemoreflex sensitivity (CHRS) is assessed in patients with stage 3 CKD [glomerular filtration rate (GFR) 30-59 ml/min/1.73 m2], in patients with stage 4 CKD [GFR 15-29 ml/min/1.73 m2], as well as in patients without any evidence of CKD. CHRS is measured by determination of the venous partial pressure of oxygen and the heart rate before and after deactivation of the chemoreceptors by inhalation of pure oxygen. The difference in the R-R intervals before and after inhalation divided by the difference in the oxygen pressures is calculated as the CHRS. A CHRS below 3.0 ms/mmHg is defined as pathological. It should be shown that using a simple clinical bedside test we provide the first evidence for impaired hyperoxic chemoreflex sensitivity in stage 3 and 4 chronic kidney disease. We thereby may lay the basis for future intervention studies assessing chemosensor function in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from CDK stage 3 (GFR 30-59 ml/min/1.73 m²) or stage 4 (GFR 15-29 ml/min/1.73 m²)
* For the reference Patients without evidence for CDK

Exclusion Criteria:

* Patients with heart failure, history of myocardial infarction or instable angina pectoris, atrial fibrillation, hyperthyroidism, chronic pulmonary diseases, sleep apnoea syndrome, alcohol abuse and drug induced cardiomyopathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Hyperoxic chemoreflex sensitivity is impaired in patients with moderate to severe chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, MD, Principal Investigator — RWTH Aachen University Departement of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonology and Vascular Medicine, Aachen, North Rhine-Westphalia, Germany